CLINICAL TRIAL: NCT06968650
Title: Efficacy of a Culturally-sensitive Telehealth Platform in Fostering Community-based Care Coordination for Respectful Maternal Care
Brief Title: Cocooned Moms Study
Acronym: Cocooned Moms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InovCares Connected Comprehensive Healthcare Corporation (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20240737; R41NR021628-01 (NIH)
Record Dates: First submitted 2025-04-25; First posted 2025-05-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Stress; Depression; Pregnancy; Blood Pressure
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- InoVCares App use (Experimental): InovCares is a culturally-sensitive telehealth platform designed for community-based care coordination in maternal care. It also offers a culturally tailored maternal mental health program, which provides access to resources addressing social determinants of health, cognitive behavioral therapy (CBT), interpersonal therapy, and compassion-focused therapy (CFT), along with peer-to-peer support and gamification. The study will evaluate the impact of these interventions on reported stress levels, depressive symptoms, sleep quality, and blood pressure (BP) among Black pregnant women
  Interventions: Behavioral: Digital and Coordinated Maternial Care

INTERVENTIONS:
Behavioral: Digital and Coordinated Maternial Care — The Cocooned Moms Study is a pre- and post-design study primarily aimed at reducing stress, depressive symptoms, and blood pressure among expectant Black women by providing them with free access to the InovCares mobile app. InovCares is a culturally-sensitive telehealth platform designed for community-based care coordination in maternal care. It also offers a culturally tailored maternal mental health program, which provides access to resources addressing social determinants of health, cognitive behavioral therapy (CBT), interpersonal therapy, and compassion-focused therapy (CFT), along with peer-to-peer support and gamification. The study will evaluate the impact of these interventions on reported stress levels, depressive symptoms, sleep quality, and blood pressure (BP) among Black pregnant women.

SUMMARY:
The Cocooned Moms Study is a pre- and post-design study primarily aimed at reducing stress, depressive symptoms, and blood pressure among expectant Black women by providing them with free access to the InovCares mobile app. InovCares is a culturally-sensitive telehealth platform designed for community-based care coordination in maternal care. It also offers a culturally tailored maternal mental health program, which provides access to resources addressing social determinants of health, cognitive behavioral therapy (CBT), interpersonal therapy, and compassion-focused therapy (CFT), along with peer-to-peer support and gamification. The study will evaluate the impact of these interventions on reported stress levels, depressive symptoms, sleep quality, and blood pressure (BP) among Black pregnant women.

ELIGIBILITY:
Inclusion Criteria:

- Black Women ages 18 + with confirmed pregnancy of at least eight or up to 28 weeks, with no known fetal or genetic abnormalities (with the exception of abnormal amniotic fluid volume; Women who have the developmental or legal capacity to consent; Able to speak English

Exclusion Criteria:

* Exclusion criteria

  1. Psychosis diagnosis
  2. Does not speak or understand English
  3. Participants who are not pregnant
  4. Non-Black
  5. Significant vision impairment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-Indentified Black Female
Enrollment: 384 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in depression, anxiety, and stress as measured by Depression Anxiety Stress Scales- Short Form (DASS-21) | Up to 7 months
  The DASS-21 at 21-items self-report measure designed to assess the severity of general psychological distress and symptoms related to depression, anxiety, and stress in adults and older adolescents. The DASS adopts a dimensional approach to psychopathology, emphasizing the degree of symptom severity rather than using diagnostic cut-offs. The overall DASS-21 score provides an indication of general psychological distress.
  Stress Subscale: The stress subscale of the DASS-21 assesses symptoms such as difficulty relaxing, nervous arousal, and being easily upset or agitated, irritable, over-reactive, or impatient. Anxiety Subscale: The anxiety subscale evaluates symptoms including autonomic arousal, effects on skeletal muscles, situational anxiety, and the subjective experience of anxious affect
Pittsburgh Sleep Quality Index (PSQI) | Up to 7 months
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month interval.
  It is frequently employed in both clinical and research settings to evaluate various aspects of sleep. The PSQI captures multiple dimensions of sleep, incorporating both subjective experiences and objective parameters. Each of the seven component scores ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The component scores are summed to produce a global PSQI score, which ranges from 0 to 21, with higher scores indicating poorer sleep quality. A score greater than 5 suggests significant sleep difficulties

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University Of Miami, Miami, Florida
  - Dr.Traci's House, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeNicola N, Grossman D, Marko K, Sonalkar S, Butler Tobah YS, Ganju N, Witkop CT, Henderson JT, Butler JL, Lowery C. Telehealth Interventions to Improve Obstetric and Gynecologic Health Outcomes: A Systematic Review. Obstet Gynecol. 2020 Feb;135(2):371-382. doi: 10.1097/AOG.0000000000003646. PMID 31977782
- [Background] Blanc J, Scaramutti C, Carrasco M, Dimanche S, Hollimon L, Moore J, Moise R, Gabbay V, Seixas A. I am Lifted Above the World: utilizing VR for stress reduction among perinatal women of color. Front Psychiatry. 2024 Apr 23;15:1377978. doi: 10.3389/fpsyt.2024.1377978. eCollection 2024. PMID 38716116
- See also: NIH Reporter — https://reporter.nih.gov/search/z4cbsZQqzUqIS2QbptonSg/projects